CLINICAL TRIAL: NCT00009048
Title: Effect of Serotoninergic Treatment in Parkinson's Disease
Brief Title: EMD 128130 for the Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010071; 01-N-0071
Record Dates: First submitted 2001-01-23; First posted 2001-01-24 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-12

CONDITIONS: Parkinson's Disease
Keywords: Dyskinesias; L-Dopa Infusion; Clinical Trial; Motor Function; Psychosis; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Dyskinesias; Psychotic Disorders | interventions — Levodopa

INTERVENTIONS:
Drug: EMD 128130
Drug: IV Levodopa

SUMMARY:
This study will evaluate the effects of an experimental drug called EMD 128130 on Parkinson's disease symptoms and on dyskinesias (involuntary movements) that develop as a result of long-term treatment with levodopa. EMD 128130 inhibits the function of serotonin, a chemical messenger thought to regulate dopamine release, and thus affect Parkinson's disease symptoms.

Patients with relatively advanced Parkinson's disease between 30 and 80 years of age may be eligible for this 3-phase study.

* Phase 1 - Baseline Evaluation

Participants will have a medical history, physical examination, detailed neurologic evaluation, routine blood tests, urinalysis and an electrocardiogram. A chest X-ray and MRI or CT scan of the brain will be done if needed. In addition, an ACTH stimulation test will be done before and at the end of the study. For this test, a hormone called ACTH is injected into a vein. A small amount of blood is drawn before the injection and 30 and 60 minutes afterwards to measure levels of another hormone called cortisol. After these tests are completed, patients will, if possible, stop taking all antiparkinsonian medications except levodopa (Sinemet) for one month before the study begins and throughout its duration.

* Phase 2 - Levodopa and Apomorphine Dose Finding

For 1 to 3 days, patients will be admitted to the NIH Clinical center to undergo a levodopa and apomorphine (a dopamine agonist) "dose-finding" procedure. For this procedure, patients will stop taking Sinemet and instead will have levodopa, and subsequently apomorphine, infused through a vein. During the infusions, the drug dose will be increased slowly until either 1) parkinsonian symptoms improve, 2) unacceptable side effects occur, or 3) the maximum study dose is reached. Symptoms will be monitored frequently to find two infusion rates: 1) one that is less than what is needed to relieve symptoms, and 2) one that relieves symptoms but may produce dyskinesias.

* Phase 3 - Active Study

Patients will begin the treatment phase within 3 months of the dose-finding phase. After a brief physical examination, routine blood tests, and evaluation of parkinsonism symptoms, patients will begin taking either EMD 128130 tablets or capsules or a placebo (a look-alike pill with no active ingredient) twice a day, along with Sinemet, for 3 weeks. All participants will receive placebo at least 1 week during the study, and about four patients, selected at random, will receive only placebo the entire 3 weeks. Levodopa and apomorphine infusions will be repeated at the end of weeks 1, 2 and 3 of Phase 3. The procedure for the infusions will be the same as in the dose-finding phase.

Throughout the study, parkinsonian symptoms and dyskinesias will be assessed and blood samples will be drawn periodically to measure drug levels. Patients will return for a follow-up evaluation 2 weeks after the end of the study.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the acute effects of a selective agonist of serotonin 5-HT1A receptors on the severity of parkinsonian signs and levodopa-associated motor response complications in patients with moderately advanced Parkinson's disease. In a controlled proof-of-principle clinical trial, the efficacy of EMD 128130 will be assessed through the use of validated motor function scales. Safety will be monitored by means of frequent clinical evaluations and laboratory tests.

ELIGIBILITY:
Males and females between the ages of 30-80.

Females must be either at least one year post-menopausal, or using an adequate contraceptive method for at least one month prior to and during participation in this study.

Patients will carry the diagnosis of idiopathic Parkinson's disease based on the presence of a characteristic clinical history and neurologic findings.

Patients will have relatively advanced disease with levodopa-associated motor response complications, including peak-dose dyskinesias and wearing-off fluctuations.

Patients with the presence or history of any medical condition that can reasonably be expected to subject the patient to unwarranted risk will be excluded.

Patients with clinically significant laboratory abnormalities including liver enzyme elevations more than two times the upper limit of normal will be excluded.

Patients who are unable to be treated with levodopa/carbidopa alone or with a single, relatively short-acting dopamine agonist will be excluded.

Patients with a form of parkinsonism other than idiopathic PD will be excluded.

Patients with unacceptable prior/concomitant medications will be excluded.

No pregnant women. Female and male patients must be practicing effective means of birth control.

Patients with prior bilateral surgical intervention for the treatment of parkinsonian symptoms, i.e. deep brain stimulation, pallidotomy, fetal tissue transplantation will be excluded.

Patients at risk for hypotension, cardiac arrhythmia, and/or myocardial ischemia secondary to intravenous levodopa challenge will not be eligible.

Patients with cognitive impairment (MMSE less than 25) will not be eligible.

Patients with subnormal serum cortisol responses to acute ACTH stimulation will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2001-01; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bernheimer H, Birkmayer W, Hornykiewicz O, Jellinger K, Seitelberger F. Brain dopamine and the syndromes of Parkinson and Huntington. Clinical, morphological and neurochemical correlations. J Neurol Sci. 1973 Dec;20(4):415-55. doi: 10.1016/0022-510x(73)90175-5. No abstract available. PMID 4272516
- [Background] Mizuno Y, Mori H, Kondo T. Parkinson's disease: from etiology to treatment. Intern Med. 1995 Nov;34(11):1045-54. doi: 10.2169/internalmedicine.34.1045. PMID 8774962
- [Background] Chase TN, Oh JD, Blanchet PJ. Neostriatal mechanisms in Parkinson's disease. Neurology. 1998 Aug;51(2 Suppl 2):S30-5. doi: 10.1212/wnl.51.2_suppl_2.s30. PMID 9711978